CLINICAL TRIAL: NCT03947203
Title: Oral Health Promotion: Youth as Agents Of Change
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to staff the project
Sponsor: Virginia Commonwealth University (Other)
Collaborators: DentaQuest Institute, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HM20014618
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Oral Hygiene
MeSH Terms: interventions — Media Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pamphlet (No Intervention): Provided with only a pamphlet containing educational material about oral health
- Social media (Experimental): Provided pamphlet containing educational material about oral health and will have access to a private Facebook group, where we will share informational messages and content relating to oral health
  Interventions: Behavioral: Social media

INTERVENTIONS:
Behavioral: Social media — Provided pamphlet and a private Facebook group where informational messages and content relating to oral health will be shared
  Arms: Social media

SUMMARY:
This upstream communication study may aid in our understanding of the nature of the parent-adolescent relationship and how we can use this relationship to promote better oral health of the parents and adolescents.

DETAILED DESCRIPTION:
Given the proliferation of social media as a tool for health communication, this proposed pilot study will be conducted with adolescents and their parents in the greater Richmond area, including Petersburg, and examines whether disseminating oral health information to adolescents via Facebook will have a greater impact on their sharing of the message to their parents than providing them the information in written format- using a pamphlet. We hypothesize that parents in the Facebook arm of the intervention will be more likely to report receiving the oral health message from their child than those in the pamphlet arm. Further, this study investigates whether parents whose adolescents re provided the information via Facebook will have greater increase in intent to schedule dental appointments and dental appointment scheduling behaviors than parents whose children are in the pamphlet group. We hypothesize that parents in the Facebook group will report greater increase in dental appointment scheduling than those whose adolescents are in the pamphlet group. Lastly, we would like to explore whether parents and adolescents in the Facebook arm will have greater increase in oral health knowledge and greater decreases in perceived barriers to oral health activities, both which may be related to increases in parents' dental appointment scheduling.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in grades 7 through 12
* between the ages of 12 and 18
* currently living in the same household as their legal guardian(s) who agree to participate in this study
* live in the greater Richmond and Petersburg area
* uses a smartphone
* has not had a dental appointment in the past 6 months

Exclusion Criteria:

* not between the ages of 12 and 18
* do not live with their legal guardian (s)
* are not residents of the greater Richmond and Petersburg area
* have had a dental appointment in the past six months
* legal guardian does not agree to participate

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Communication | 8 weeks
  Sharing of health information measured as a count of shared oral health messages reported on a survey question.
Appointment - child | 8 weeks
  Number of child dental appointments scheduled based on self-report
Appointment - adult | 8 weeks
  Number of adult dental appointments scheduled based on self-report

SECONDARY OUTCOMES:
Oral health knowledge | Baseline to 8 weeks
  Change in number of correct responses on a 12 item oral health knowledge and screening survey
Perceived barriers | Baseline to 8 weeks
  Change in number of barriers to oral health activities

CONTACTS AND LOCATIONS:
Overall Officials: Maghboobah Mosavel, MD, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No